CLINICAL TRIAL: NCT03536052
Title: Ablation at Virtual-hEart pRedicted Targets for VT
Acronym: AVERT-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00141401
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Virtual Heart Guided Ablation (Experimental)
  Interventions: Device: Virtual Heart Guided Ablation

INTERVENTIONS:
Device: Virtual Heart Guided Ablation — If a good quality cardiac MRI is obtained and a virtual heart model with the ablation targets is generated, the operating physician will merge the virtual heart lesion map to the invasive electroanatomical navigation system. After the patient has been catheterized, an attempt should be made to induce VT. The physician should then navigate the catheter to each of the ablation targets specified, and place a lesion as per his or her training and experience, confirming when done that the lesion marker in the mapping system coincides with the target. This will be done for each lesion.

SUMMARY:
The goal of this study is to test the efficacy of the new imaging/simulation ("virtual heart") approach for determining the optimal ablation sites in patients with VT, which render post-infarction VT non-inducible. The study will test both the acute outcome of the ablation procedure, and the effect the use of the predicted targets has upon procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must be at least 18 years old at the time of enrollment.
* A Pre-Op cardiac MRI including late gadolinium enhancement (LGE) must be performed prior to ablation. As Johns Hopkins University (JHU) performs MRIs with implantable cardioverter defibrillator (ICD) or pacemaker implanted, patients with these devices may be enrolled.
* Eligible patients must suffer from VT, thought to be secondary to structural heart disease (scarring).
* Eligible patients must be determined to be suitable candidates for ablation to treat VT by their cardiologist and/or electrophysiologists regardless of this protocol.

Exclusion Criteria:

* Patients with Glomerular Filtration Rate (GFR) < 30 mL/min should not be enrolled in the study due to the use of intravenous gadolinium as an MRI contrast agent
* If a pre-procedure MRI cannot or likely will not be performed for any reason (such as claustrophobia), the patient must be excluded.
* Pregnant women may not participate in the study because gadolinium MRI contrast is contraindicated in these patients.
* Any subject that, during the course of the pre-procedure imaging, is discovered to have VT not related to scarring, he/she must be de-enrolled from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chrispin, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Heart Guided Ablation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Virtual Heart Guided Ablation: Participants undergoing Virtual Heart Guided Ablation
Arm/Group | Virtual Heart Guided Ablation
Number analyzed (Participants) | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 70.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ventricular Tachycardia Inducibility
Description: Following ablation, inducibility of VT will be determined using programmed electrical stimulation
Time Frame: time of procedure
Population: 3 participatnts were not included in the primary analysis. 2 participants were not inducible for ventricular tachycardia at the beginning of the procedure. 1 participant was not hemodynamically stable to attempt re induction of ventricular tachycardia
Measure: Count of Participants; unit: Participants
Groups:
- Virtual Heart Guided Ablation: Participants undergoing virtual heart-guided ablation
Arm/Group | Virtual Heart Guided Ablation
Number analyzed (Participants) | 7
Participants | 6

2. Secondary Outcome: Freedom From Ventricular Tachycardia
Description: Long term Freedom of Spontaneous Ventricular Tachycardia
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Heart Guided Ablation
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 1 year
Groups:
- Virtual Heart Guided Ablation: Participant undergoing virtual heart-guided ablation
Arm/Group | Virtual Heart Guided Ablation
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT03536052/Prot_003.pdf